CLINICAL TRIAL: NCT04270565
Title: Gait-Training Using Wearable Sensors for Runners With Exercise-Related Lower Leg Pain
Brief Title: Gait-Training Using Wearable Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jay Hertel, PhD, ATC, Joe H. Gieck Professor of Sports Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22107
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Shin Splint; Running-related Injury
Keywords: running; gait-training; exercise-related lower leg pain; wearable sensors
MeSH Terms: conditions — Medial Tibial Stress Syndrome

STUDY DESIGN:
Intervention Model Description: There will be two groups:
  1. real-time gait-training interventions along with a home exercise program (intervention group)
  2. only home exercise program (control group).
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The investigator assessing laboratory-based outcome measures will be blinded to group allocation. Additionally, the investigator designing the home exercise program and making progression decisions will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive real-time gait-training interventions along with a home exercise program. Participants in this group will be given a pair of sensors to wear on their shoes to wear during runs throughout the study period, and wear a Garmin watch to get information from the sensors to the watch for feedback. They will also do home exercises during the study, and to come into the laboratory weekly for about 30 minutes per visit to progress the home exercises and get instructions on feedback for the next week.
  Interventions: Behavioral: In-Field Gait-Training; Behavioral: Home Exercise
- Control Group (Active Comparator): The control group will receive only a home exercise program. Participants in this group will be given a pair of sensors to wear on their shoes to wear during runs throughout the study period, and do home exercises during the study. Participants will be asked to come into the laboratory weekly for about 30 minutes per visit to progress the home exercises.
  Interventions: Behavioral: Home Exercise

INTERVENTIONS:
Behavioral: In-Field Gait-Training — The intervention will deliver a series of vibrations on the participants' wrists through the Garmin when the sensors indicate that their contact time in milliseconds exceeds a threshold. The runners will be asked to reduce the amount of time their foot is in contact with the ground by picking their feet up more quickly. Participants will also receive a series of exercises based on noted impairments at baseline. The feedback during running will be completed twice per week for four weeks.
  Other Names: RunScribe; Garmin
  Arms: Intervention Group
Behavioral: Home Exercise — Participants will receive a series of exercises based on noted impairments at baseline. Exercises will be completed twice per week for four weeks.

SUMMARY:
The overarching purpose of this project is to use sensor-derived patterns to guide running interventions during in-field training scenarios for runners with exercise-related lower leg pain. The investigators plan to use the RunScribe sensors to facilitate in-field gait-training to determine the effects of real-time gait-training interventions along with a home exercise program (intervention group) on biomechanical and patient-reported outcome measures of pain and function in runners with leg pain as opposed to receiving a home exercise program alone (control group).

DETAILED DESCRIPTION:
The purpose of the study is to determine the effects of real-time gait-training interventions along with a home exercise program (intervention group) on biomechanical and patient-reported outcome measures of pain and function in runners with leg pain as opposed to receiving a home exercise program alone (control group). All participants will report to the Exercise and Sport Injury Laboratory for a 60-minute baseline clinical assessment performed by a blinded assessor to determine hip, knee, foot and ankle strength, range of motion, and alignment using valid and reliable measurement techniques. Participants will also perform a series of functional movement assessments while an assessor records frontal and sagittal camera views in order to determine lower extremity dynamic alignment. The functional assessments will include the star excursion balance test (SEBT), a lateral step-down, a single-leg squat to 45 degrees of knee flexion, and a treadmill gait assessment. The movement screens will be use to form criteria-based home exercise programs, such that a blinded assessor will evaluate the videos and categorize patients into varus, valgus, or neutral alignment groups. Participants will receive exercises tailored to these descriptions. Further, the static alignment measurements will be used to determine if lower extremity stretches are warranted.

Following the first baseline visit, participants will return to the lab for a second baseline visit to complete an indoor, instrumented gait analysis using a motion capture system. Participants will also become oriented to the RunScribe wearable sensors and associated phone application, and will perform a brief outdoor run at their preferred speed to calibrate the sensors. Participants will receive their home exercise prescription with supplemental videos to take home with them to ensure adequate understanding of the target exercise performance. Participants will then be randomly assigned to one of two groups: 1) sensor-based feedback with home exercises (intervention group), or 2) home exercises alone (control group). The randomization sequence will be created a priori with a random-number generator stratified by sex, and allocation will be placed in a sealed opaque envelope by the graduate student mentor to intentionally blind the study coordinator conducting the interventions.

Participants in the intervention group will receive a Garmin wristwatch to facilitate the gait-training feedback, and will be oriented to the procedures during 10 minutes of running on an indoor treadmill in the presence of the study coordinator to ensure adequate understanding and integration of the feedback. The RunScribe sensors will facilitate the feedback by providing real-time metrics on the Garmin watch face using a custom application. Contact time will be the central focus of the intervention; participants will receive a vibro-tactile alert to remain below the identified contact time cut-off based on preliminary data.

Regardless of group allocation, participants will be instructed to maintain a running log within the RunScribe phone application to track activity adherence, details of runs that are recorded by the sensors, and report pain 1-10 experienced before, during, and after runs. All participants will be asked to perform their interventions twice per week. Participants will be encouraged to maintain other normal activities in addition to the interventions.

During the intervention period, all participants will return to the lab once per week to determine if exercise progressions are warranted based using specific performance-based scoring criteria. These decisions will be made by an assessor blinded to group allocation. The intervention group participants will then check in with the unblinded study coordinator to receive instructions on gait-training feedback progressions. The intervention will follow a volume-based faded feedback design.

At the midpoint of the study, all participants will complete Visual Analog and Global Rating of Change scales to track self-reported recovery. At the end of the intervention period, all participants will be re-assessed by the same blinded assessor using the same baseline measures to determine changes in lower limb alignment, strength, flexibility, and functional movement patterns. The indoor gait assessment and calibration run performed at the second baseline visit will be repeated at this follow-up timepoint while all participants wear the RunScribe sensors. Participants will also repeat Visual Analog Pain and Global Rating of Change scales to assess self-reported recovery. The investigators will then be able to determine if contact time feedback delivered in the field effectively decreases contact time after feedback compared to baseline and compared to the control group, determine if contact time feedback delivered in the field carries over to other gait outcomes in the intervention group after gait-training compared to baseline and the control group, and assess if pain decreases and function increases after gait-training compared to baseline and to a greater extent than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45 years
* Male or female
* Involved in running training at least two times per week over the past three months
* Current weekly mileage of at least 6 miles
* Currently experiencing pain during or after running in the anterior or medial aspect of the leg (between the knee and the ankle) of at least one week in duration, with maximum pain levels between 3/10 and 8/10 on the Visual Analogue Scale
* All subjects must be willing to use their own smart phone device (iPhone or Android) to download the RunScribe application for study procedures.

Exclusion Criteria:

* Primary complaint is of pain over the Achilles tendon, popliteal fossa, or lateral or superficial posterior compartment of the lower leg
* Medical diagnosis of compartment syndrome, tibial or fibular stress fracture, or tibial or fibular fracture within the past 3 months
* Current running-related injuries within 3 months at the foot, ankle, knee, thigh, hip, or lower back
* Any history of lower extremity or lower back surgery
* Subjects with known pregnancy
* Subject with any type of neuropathy (numbness/tingling) in lower extremity
* Subject with clinical diagnosis of Parkinson's disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Contact Time | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  the amount of time (in milliseconds) the foot is in contact with the ground as measured using the RunScribe sensors
Change in Contact Time Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  the amount of time (in milliseconds) the foot is in contact with the ground as measured using the RunScribe sensors
Maintaining Change in Contact Time | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  the amount of time (in milliseconds) the foot is in contact with the ground as measured using the RunScribe sensors
Change in Hip Frontal Plane Motion | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Hip frontal plane motion (in degrees) measured during the indoor motion capture gait analysis on a treadmill
Change in Gluteus Medius Electromyography | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Normalized gluteus medius muscle activity root mean square electromyography measured during the indoor motion capture gait analysis on a treadmill
Change in Tibialis Anterior Electromyography | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Normalized tibialis anterior muscle activity root mean square electromyography measured during the indoor motion capture gait analysis on a treadmill
Change in Pain Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Visual Analog Scale (0-100 mm) pain outcome scores
Maintaining Change in Pain Outcomes | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  Visual Analog Scale (0-100 mm) pain outcome scores
Maintaining Change in Exercise-Induced Leg Pain Questionnaire - British Version Outcomes | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  Exercise Induced Leg Pain Questionnaire - British Version (0-100%) outcome scores
Change in Pain Outcomes Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  Visual Analog Scale (0-100 mm) pain outcome scores
Change in Exercise-Induced Leg Pain Questionnaire - British Version Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Exercise Induced Leg Pain Questionnaire - British Version (0-100%) outcome scores
Change in Step Rate | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  the step rate per minute (in steps/min) during running as measured using the RunScribe sensors
Change in Stride Length | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  the distance the legs reach out (in meters) during running as measured using the RunScribe sensors
Change in Maximum Pronation Velocity | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  the speed in which the foot turns over, or pronates, (in degrees/sec) during running as measured using the RunScribe sensors
Change in Shock | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  the extent of lower extremity loading (in g's) during running as measured using the RunScribe sensors
Change in Foot Strike Type | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  the area on the foot that participants land on (on a 1-16 scale, with 1 indicating rear foot strike and 16 indicating a forefoot strike) during running as measured using the RunScribe sensors
Change in Exercise-Induced Leg Pain Questionnaire - British Version Outcomes Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  Exercise Induced Leg Pain Questionnaire - British Version (0-100%) outcome scores

SECONDARY OUTCOMES:
Change in Peroneus Longus Electromyography | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Normalized peroneus longus muscle activity root mean square electromyography measured during the indoor motion capture gait analysis on a treadmill
Change in Medial Gastocnemius Electromyography | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Normalized medial gastrocnemius muscle activity root mean square electromyography measured during the indoor motion capture gait analysis on a treadmill
Change in Foot Strike Type Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  the area on the foot that participants land on (on a 1-16 scale, with 1 indicating rear foot strike and 16 indicating a forefoot strike) during running as measured using the RunScribe sensors
Change in Shock Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  the extent of lower extremity loading (in g's) during running as measured using the RunScribe sensors
Change in Maximum Pronation Velocity Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  the speed in which the foot turns over, or pronates, (in degrees/sec) during running as measured using the RunScribe sensors
Change in Stride Length Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  the distance the legs reach out (in meters) during running as measured using the RunScribe sensors
Change in Step Rate Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  the step rate per minute (in steps/min) during running as measured using the RunScribe sensors
Maintaining Change in Foot Strike Type | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  the area on the foot that participants land on (on a 1-16 scale, with 1 indicating rear foot strike and 16 indicating a forefoot strike) during running as measured using the RunScribe sensors
Maintaining Change in Shock | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  the extent of lower extremity loading (in g's) during running as measured using the RunScribe sensors
Maintaining Change in Maximum Pronation Velocity | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  the speed in which the foot turns over, or pronates, (in degrees/sec) during running as measured using the RunScribe sensors
Maintaining Change in Stride Length | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  the distance the legs reach out (in meters) during running as measured using the RunScribe sensors
Maintaining Change in Step Rate | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  the step rate per minute (in steps/min) during running as measured using the RunScribe sensors
Change in Hip Sagittal Plane Motion | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Hip sagittal plane motion (in degrees) measured during the indoor motion capture gait analysis on a treadmill
Change in Hip Sagittal Plane Kinetics | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Hip sagittal plane joint moment (in Nm/kg) measured during the indoor motion capture gait analysis on a treadmill
Change in Hip Transverse Plane Motion | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Hip transverse plane motion (in degrees) measured during the indoor motion capture gait analysis on a treadmill
Change in Hip Transverse Plane Kinetics | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Hip transverse plane joint moment (in Nm/kg) measured during the indoor motion capture gait analysis on a treadmill
Change in Hip Frontal Plane Kinetics | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Hip frontal plane joint moment (in Nm/kg) measured during the indoor motion capture gait analysis on a treadmill
Change in Knee Frontal Plane Motion | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Knee frontal plane motion (in degrees) measured during the indoor motion capture gait analysis on a treadmill
Change in Knee Frontal Plane Kinetics | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Knee frontal plane joint moment (in Nm/kg) measured during the indoor motion capture gait analysis on a treadmill
Change in Knee Sagittal Plane Kinetics | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Knee sagittal plane joint moment (in Nm/kg) measured during the indoor motion capture gait analysis on a treadmill
Change in Ankle Sagittal Plane Motion | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Ankle sagittal plane motion (in degrees) measured during the indoor motion capture gait analysis on a treadmill
Change in Ankle Sagittal Plane Kinetics | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Ankle sagittal plane joint moment (in Nm/kg) measured during the indoor motion capture gait analysis on a treadmill
Change in Knee Sagittal Plane Motion | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Knee sagittal plane motion (in degrees) measured during the indoor motion capture gait analysis on a treadmill
Change in Trunk Frontal Plane Motion | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Trunk frontal plane motion (in degrees) measured during the indoor motion capture gait analysis on a treadmill
Change in Trunk Sagittal Plane Motion | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Trunk sagittal plane motion (in degrees) measured during the indoor motion capture gait analysis on a treadmill
Change in Trunk Frontal Plane Kinetics | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Trunk frontal plane joint moment (in Nm/kg)measured during the indoor motion capture gait analysis on a treadmill
Change in Trunk Sagittal Plane Kinetics | This outcome change will be measured from baseline to the end of the intervention (4 weeks) for both groups.
  Trunk sagittal plane joint moment (in Nm/kg) measured during the indoor motion capture gait analysis on a treadmill
Maintaining Global Change Outcomes | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  Global Rating of Change Scale (11-point scale)
Maintaining Recovery Outcomes | This outcome change will be assessed from the end of the intervention (4 weeks) to follow-up at 6 weeks for both groups.
  Wisconsin Injury and Recovery Scale (0-100%)
Change in Recovery Outcomes Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  Wisconsin Injury and Recovery Scale (0-100%)
Change in Global Change Outcomes Across the Intervention Period | This outcome change will be assessed through study completion over 4 weeks for both groups.
  Global Rating of Change Scale (11-point scale)
Change in Single-Leg Squat Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  single-leg squat to 45 degrees of knee flexion functional performance scores (valgus, varus, or neutral scoring)
Change in Lateral Step-Down Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  lateral step-down from a 35 cm box functional performance scores (valgus, varus, or neutral scoring)
Change in Star Excursion Balance Test Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  star excursion balance test performance scores (reach distances as a % of leg length for 8 reach directions)
Change in Visual Gait Analysis Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  visual gait assessment functional performance score (valgus, neutral, or varus)
Change in Foot Posture Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical foot posture index assessment (23-point scale)
Change in Arch Height Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical arch height index assessment using a Jaktool (ratio of seated to standing measures)
Change in Weight-Bearing Dorsiflexion Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical weight-bearing dorsiflexion (knee-to-wall) assessment (in centimeters)
Change in Ankle Plantarflexion Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Ankle Dorsiflexion Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Metatarsophalangeal Joint Flexion Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Metatarsophalangeal Joint Extension Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Hip Abduction Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Ankle Inversion Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Ankle Eversion Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Knee Flexion Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Tibial Torsion Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Hip Anteversion Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical range of motion assessment using standard goniometer (in degrees)
Change in Hamstring Flexibility Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing hamstring flexibility, called the 90/90 straight leg raise test (in degrees)
Change in Hip Flexor Flexibility Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing hip flexor flexibility, called the Thomas test (in centimeters)
Change in Metatarsophalangeal Joint Flexion Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)
Change in Ankle Dorsiflexion Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)
Change in Ankle Plantarflexion Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)
Change in Ankle Inversion Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)
Change in Ankle Eversion Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)
Change in Hip Flexion Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)
Change in Hip Extension Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)
Change in Hip Abduction Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)
Change in Knee Extensor Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)
Change in Knee Flexor Strength Outcomes | This outcome change will be assessed from baseline to the end of the intervention (4 weeks) for both groups.
  Clinical test assessing strength using hand-held dynamometry (in N/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hertel, PhD, Principal Investigator — University of Virginia
Locations (1):
- Memorial Gymnasium - Exercise and Sport Injury Laboratory, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willy RW. Innovations and pitfalls in the use of wearable devices in the prevention and rehabilitation of running related injuries. Phys Ther Sport. 2018 Jan;29:26-33. doi: 10.1016/j.ptsp.2017.10.003. Epub 2017 Oct 6. PMID 29172095
- [Background] Koldenhoven RM, Hertel J. Validation of a Wearable Sensor for Measuring Running Biomechanics. Digit Biomark. 2018 Aug 2;2(2):74-78. doi: 10.1159/000491645. eCollection 2018 May-Aug. PMID 32095758
- [Background] Hollis CR, Koldenhoven RM, Resch JE, Hertel J. Running biomechanics as measured by wearable sensors: effects of speed and surface. Sports Biomech. 2021 Aug;20(5):521-531. doi: 10.1080/14763141.2019.1579366. Epub 2019 Mar 7. PMID 30843475
- [Background] DeJong AF, Hertel J. Gait-training devices in the treatment of lower extremity injuries in sports medicine: current status and future prospects. Expert Rev Med Devices. 2018 Dec;15(12):891-909. doi: 10.1080/17434440.2018.1551130. Epub 2018 Dec 10. PMID 30466335
- [Background] Willems TM, Witvrouw E, De Cock A, De Clercq D. Gait-related risk factors for exercise-related lower-leg pain during shod running. Med Sci Sports Exerc. 2007 Feb;39(2):330-9. doi: 10.1249/01.mss.0000247001.94470.21. PMID 17277598
- [Background] Reinking MF, Hayes AM. Intrinsic factors associated with exercise-related leg pain in collegiate cross-country runners. Clin J Sport Med. 2006 Jan;16(1):10-4. doi: 10.1097/01.jsm.0000188041.04760.d2. PMID 16377969
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Korakakis V, Malliaropoulos N, Baliotis K, Papadopoulou S, Padhiar N, Nauck T, Lohrer H. Cross-cultural Adaptation and Validation of the Exercise-Induced Leg Pain Questionnaire for English- and Greek-Speaking Individuals. J Orthop Sports Phys Ther. 2015 Jun;45(6):485-96. doi: 10.2519/jospt.2015.5428. Epub 2015 Apr 30. PMID 25927499
- [Background] Abbott JH, Wright AA. Global Rating of Change (GROC): the minimally important change at which patients choose to stop seeking treatment. N Z J Physiother. 2010;38(2):66-66.
- [Background] Nelson EO, Ryan M, AufderHeide E, Heiderscheit B. Development of the University of Wisconsin Running Injury and Recovery Index. J Orthop Sports Phys Ther. 2019 Oct;49(10):751-760. doi: 10.2519/jospt.2019.8868. Epub 2019 Aug 3. PMID 31378123
- [Derived] DeJong Lempke AF, Stephens SL, Fish PN, Thompson XD, Hart JM, Hryvniak DJ, Rodu JS, Hertel J. Sensor-based gait training to reduce contact time for runners with exercise-related lower leg pain: a randomised controlled trial. BMJ Open Sport Exerc Med. 2022 Nov 3;8(4):e001293. doi: 10.1136/bmjsem-2021-001293. eCollection 2022. PMID 36353183